CLINICAL TRIAL: NCT02394860
Title: Influence of Periodontal Diseases on Hemodynamic and Molecular Vascular Parameters in Patients Suffering of Hypertension
Brief Title: Influence of Periodontal Diseases on Vascular Parameters in Patients Suffering of Hypertension
Status: Terminated | Type: Observational
Why Stopped: no patient
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5883
Record Dates: First submitted 2014-07-08; First posted 2015-03-20 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Periodontitis; Hypertension
MeSH Terms: conditions — Chronic Periodontitis; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- blood and cardiological examination
  Interventions: Other: echo Doppler lower limbs

INTERVENTIONS:
Other: echo Doppler lower limbs

SUMMARY:
The aim of this study is to assess the influence of the severity of chronic periodontitis on hemodynamic parameters in hypertensive patients.Secondary purposes of this protocol is to identify evolution of several biomarkers and correlate the clinical situation with oral microflora.

ELIGIBILITY:
Inclusion Criteria:

* -Men- >40 years
* moderate and severe generalized chronic periodontitis
* Former diagnosis of hypertension
* >12 teeth

Exclusion Criteria:

* >70 years
* smokers (>10 cig/day)
* body mass index>30
* Need of antibioprophylaxis
* Medical treatment including anti-inflammatory drugs and/or antibiotics
* Refractory form of hypertension- aggressive periodontitis

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will be included men with severe and moderate periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2024-02 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Measuring the thickness of the intima-media | 15 days

SECONDARY OUTCOMES:
Evaluation of anatomical changes that may occur at the arterial level | Within 15 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HUCK, MD, Principal Investigator — CHRU Strasbourg
Locations (1):
- Service de parodontologie, Strasbourg, France